CLINICAL TRIAL: NCT00759447
Title: A Multicenter Pilot Study to Evaluate the Image Quality of Two Hologic Tomosynthesis Mammography Systems
Brief Title: A Pilot Study - Comparison of Two Hologic 3D Mammography Systems
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-01
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- 3D investigational imaging: Patients enrolled will be imaged with a 3D mammogram in one of 3 speeds of acquisition
  Interventions: Device: Investigational 3D Mammography system
- 3D Imaging with commercial Mammography Device
  Interventions: Device: Genesis and Gemini

INTERVENTIONS:
Device: Genesis and Gemini — 3 dimensional breast mammography system
  Other Names: Selenia Dimensions
  Groups: 3D Imaging with commercial Mammography Device
Device: Investigational 3D Mammography system — 3 dimensional breast mammography system
  Groups: 3D investigational imaging

SUMMARY:
Study to compare the prototype tomosynthesis mammography system to the tomosynthesis system slated for commercial release.

DETAILED DESCRIPTION:
A perspective non randomized, noncontrolled, multicenter pilot study enrolling a minimum of 60 female subjects. The purpose of the pilot study is to compare the images acquired from two Hologic tomosynthesis systems. Information obtained from the study will be used to determine endpoints for a future larger study. Study participants are enrolled in one of three groups, the group in which they are enrolled wil determine which tomosynthesis system images will be acquired upon.

ELIGIBILITY:
Inclusion Criteria:

* Female, any ethnic origin
* No contraindication for diagnostic mammography

Exclusion Criteria:

* Any contraindications to mammographic imaging including but not limited to significant existing breast trauma, pregnancy, lactating, breast implants.
* Under 30 years of age at the time of consent
* Unable to understand and execute written informed consent

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female who are undergoing screening mammography.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pilot study- To Evaluate the images acquired on 2 prototype systems for a larger study design | 1 year
  images are acquired on 2 systems with different speeds of time and reviewed compared to 2D images. Subjects are enrolled in one group or another and are diagnostic patients returning for addition work up on an area of interest